CLINICAL TRIAL: NCT03715660
Title: Xpert Bladder Cancer Monitor; Prospective, Single, Tertiary-care Center Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE 2395
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Bladder Cancer
Keywords: Non muscle invasive bladder cancer, recurrence, progression
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Recurrence; Disease Progression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xpert monitor- evaluated patients (Experimental): Xpert Bladder Cancer Monitor performance shall be established in recurrence patients relative to cystoscopy (for disease negative patients) or histology (for disease positive patients)and relative to a currently used diagnostic assay (urine cytology)which is the standard of care used for detecting recurrent bladder cancer at the site. In this study, clinical sensitivity shall be established in patients who have been previously diagnosed with bladder cancer and are scheduled for a standard of care (SOC) surveillance cystoscopy.
  Interventions: Diagnostic Test: Xpert bladder cancer monitor

INTERVENTIONS:
Diagnostic Test: Xpert bladder cancer monitor — Xpert Bladder Cancer Monitor, is a qualitative in vitro diagnostic test designed to monitor for the recurrence of bladder cancer in patients previously diagnosed with bladder cancer.The test utilizes a voided urine specimen and measures the levels of five targetmRNAs (ABL1, CRH, IGF2, UPK1B, ANXA10) by means of real-time, reverse transcription-polymerase chain reaction (RT-PCR). The Xpert Bladder Cancer Monitor is indicated as an aid to standard clinical evaluation in monitoring for bladder cancer recurrence in patients previously diagnosed with bladder cancer and should be used in conjunction with other clinical measures to assess disease recurrence.

SUMMARY:
The primary objective of this prospective, single-centre study is to establish the clinical performance characteristics of Xpert Bladder Cancer Monitor on the GeneXpert Instrument Systems in comparison to the methods currently used at the site for detecting recurrent bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient shall meet all of the following criteria in order to be considered eligible for enrollment:

  * Patient has been diagnosed with NMIBC within 24 months of enrollment
  * At the time of the enrollment visit, the patient is scheduled for a cystoscopy within the next 6 weeks of enrollment

Exclusion Criteria:

* Patient has had an excision procedure or BCG treatment within six weeks (42 days) before enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Xpert Bladder Cancer Monitor in monitoring of non muscle invasive bladder cancer by comparing its results to the results of the standard tool of monitoring of bladder cancer (diagnostic cystoscopy) | within 1 month after test assessment
  Xpert Bladder Cancer Monitor performance shall be established in recurrence patients relative to cystoscopy (for disease negative patients) or histology (for disease positive patients)and relative to a currently used diagnostic assay (urine cytology)which is the standard of care used for detecting recurrent bladder cancer at the site. In this study, clinical sensitivity shall be established in patients who have been previously diagnosed with bladder cancer and are scheduled for a standard of care (SOC) surveillance cystoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt